CLINICAL TRIAL: NCT06728176
Title: A Single Centre, Double Blinded, Randomised, Parallel Arm, Placebo Controlled Study to Evaluate the Safety and Pharmacokinetics of MT1988 in Healthy Adults
Brief Title: Safety and PK of Multiple Doses of MT1988
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Monument Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCZ103
Record Dates: First submitted 2024-12-02; First posted 2024-12-11 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteer
Keywords: Phase I

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- MT1988 Dose 1 (Experimental): MT1988 Dose Level 1 (oral, twice daily)
  Interventions: Drug: MT1988
- MT1988 Dose 2 (Experimental): MT1988 Dose Level 2 (oral, twice daily)
  Interventions: Drug: MT1988
- MT1988 Dose 3 (Experimental): MT1988 Dose Level 3 (oral, twice daily)
  Interventions: Drug: MT1988
- MT1988 Dose 4 (Experimental): MT1988 Dose Level 4 (oral, twice daily)
  Interventions: Drug: MT1988
- Placebo (Placebo Comparator): Placebo (oral, twice daily)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT1988 — Active Drug
  Arms: MT1988 Dose 1; MT1988 Dose 2; MT1988 Dose 3; MT1988 Dose 4
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the tolerability and amount of drug in the blood when four dose levels of MT1988 are administered for 14 days to healthy volunteers. The main question it aims to answer is:

* what side effects are seen while administering MT1988 for 14 days?
* how much of MT1988 can be measured in the blood at the beginning and end of administering MT1988 for 14 days?

Researchers will include a placebo arm (dummy drug) to compare the side effects.

Participants will:

* take MT1988 every day for 14 days
* visit the clinic once per week for assessments
* keep a diary to record information between clinic appointments.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* providing informed consent
* for females of child-bearing potential with fertile male partner - willing to comply with contraception requirements

Exclusion Criteria:

* no current or past condition which may compromise the study objectives or participant safety
* no clinically significant finding at screening, including physical examination, blood tests, medical history, concomitant medication
* history of drug abuse or dependence within the previous 2 years

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | From Day 1 to end of follow up (Day 21-28)
  Data will be analysed using descriptive statistics across four dose levels and versus placebo.

SECONDARY OUTCOMES:
Pharmacokinetics of single dose of MT1988 across four dose levels - Cmax | Days 1-2
  Maximum plasma concentration (Cmax). Between-group comparisons will be made using descriptive statistics
Pharmacokinetics of multiple doses of MT1988 across four dose levels - Cmax | Days 14 to 17
  Maximum plasma concentration (Cmax). Between-group comparisons will be made using descriptive statistics
Pharmacokinetics of single doses of MT1988 across four dose levels - Tmax | Days 1-2
  Time to maximum plasma concentration (Tmax). Between-group comparisons will be made using descriptive statistics
Pharmacokinetics of multiple doses of MT1988 across four dose levels - Tmax | Days 14 to 17
  Time to maximum plasma concentration (Tmax). Between-group comparisons will be made using descriptive statistics
Pharmacokinetics of single doses of MT1988 across four dose levels - AUC | Days 1-2
  Total drug exposure (area under the curve (AUC))). Between-group comparisons will be made using descriptive statistics
Pharmacokinetics of multiple doses of MT1988 across four dose levels - AUC | Days 14 to 17
  Total drug exposure (area under the curve (AUC))). Between-group comparisons will be made using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Principal Investigator — BDD Pharma
Locations (1):
- BDD Pharma Ltd, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Sharing of IPD is not appropriate for this Phase I commercial study in healthy volunteers